CLINICAL TRIAL: NCT03014219
Title: A Phase I Study of Autologous Mesenchymal Stromal Cell Coated Fistula Plug in Patients With Fistulizing Crohn's Disease: Pediatric Sub-study
Brief Title: Phase 1 Crohn's Pediatric Sub-study of MSC AFP
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA approval was not obtained until adult trial completes accrual
Sponsor: William A. Faubion, M.D. (Other)
Responsible Party: Sponsor-Investigator, William A. Faubion, M.D., Sponsor Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-005574
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Perianal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Only 1 arm: treatment with MSC-AFP (Experimental): Single Treatment Group: Eligible patients will be treated with a Gore Bio-A Fistula Plug that has been coated with autologous mesenchymal stromal cells. This is a drug study, specifically phase 1 study of autologous mesenchymal stromal cells. Single dose of 20 million cells.
  Interventions: Drug: Only 1 arm: treatment with MSC-AFP

INTERVENTIONS:
Drug: Only 1 arm: treatment with MSC-AFP — Eligible patients will be treated with a fistula plug that has been coated with autologous mesenchymal stromal cell. Drug study. Single dose of 20 million cells.
  Other Names: mesenchymal stromal cells

SUMMARY:
The investigators propose to study the safety of autologous mesenchymal stromal cell transfer using a biomatrix (the Gore Bio-A Fistula Plug) in a Phase I study using a single dose of 20 million cells. 20 patients (age 12 to 17 years) with Crohns perianal fistulas will be enrolled.

Subjects will undergo standard adjuvant therapy including drainage of infection and placement of a draining seton. Six weeks post placement of the draining seton, the seton will be replaced with the MSC loaded Gore fistula plug as per current clinical practice. The subjects will be subsequently followed for fistula response and closure for 24 months. This is an autologous product derived from the patient and used only for the same patient.

DETAILED DESCRIPTION:
Visit 1: Patients will be evaluated for eligibility (inclusion/exclusion checklist) and written, informed consent will be obtained. Patients will undergo general exam with vital signs. Patients will be scheduled for a fat biopsy to collect the tissue needed to grow MSC. In the event there is no cell growth from the tissue obtained from the first biopsy, one further attempt will made from a second tissue sample from this patient. However, if the second attempt fails to grow cells, no further attempts will be made, and the subject will not continue in the study.

The subjects will be subsequently followed for fistula response and closure for 24 months. Study visits are Day 1, Week 2, Week 4, Week 8, Week 12, Week 24, Week 52, and Week 104. This is an autologous product derived from the patient and used only for the same patient.

ELIGIBILITY:
Inclusion Criteria

1. Males and females 12-17 years of age.
2. Residents of the United States.
3. Crohn's disease with single or multiple draining complex perianal fistulae (definition as below) for at least three months despite standard therapy (definition below).
4. Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, and anti-TNF therapy are permitted.
5. All patients should have undergone a colonoscopy in last 12 months to rule out malignant or premalignant condition
6. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
7. Ability to comply with protocol
8. Competent and able to provide written informed consent (and assent where appropriate).
9. Must have failed standard medical therapy including anti-TNF agents

Exclusion Criteria

1. Inability to obtain informed consent (and assent where appropriate).
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. sepsis, pneumonia active serious infection or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
3. Specific exclusions;

   a. Evidence of hepatitis B, C, or HIV
4. History of cancer including melanoma (with the exception of localized skin cancers)
5. Investigational drug within thirty (30) days of baseline
6. A resident outside the United States
7. Pregnant or trying to become pregnant, or breast feeding.
8. History of clinically significant auto-immunity (other than Crohn's disease) or any previous example of fat-directed autoimmunity
9. Previous allergic reaction to a perianal fistula plug.
10. If adipose tissue is not technically feasible
11. Weight less than 35 kg
12. Allergic to local anesthetics
13. Non-enterocutaneous tracts (i.e. recto-vaginal, entero-vesicular)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with any Adverse Events that are related to study drug | [Time Frame: 2-24 months
  The primary endpoint of this study is to determine the safety of using adipose derived, autologous mesenchymal stromal cells (MSC) bound to the Gore Bio-A Fistula Plug for treatment of refractory CD perianal fistulae.

SECONDARY OUTCOMES:
Number of Subjects with healing in response to the study drug treatment | Time Frame: 2-24 months
  The Outcome Measure will be the presence or absence of fistula drainage (Yes vs. No)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Stephens, Principal Investigator — Mayo Clinic; William Faubion, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States